CLINICAL TRIAL: NCT01047072
Title: Phase II Clinical Trial of Allogeneic Hematopoietic Cell Transplantation After Nonmyeloablative Conditioning for Patients With Severe Systemic Sclerosis
Brief Title: Low-Dose Conditioning Followed by Donor Stem Cell Transplant in Treating Patients With Severe Systemic Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Georges, George, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2363.00; NCI-2012-00139 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Systemic Scleroderma
Keywords: Scleroderma, systemic sclerosis, allogeneic hematopoietic stem cell transplantation
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — fludarabine phosphate; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Rituximab; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (transplant) (Experimental): Patients receive fludarabine IV on days -4 to -2. Patients undergo total-body irradiation on day 0. Patients then undergo peripheral blood stem cell transplantation on day 0. Patients receive GVHD prophylaxis comprising tacrolimus PO twice daily on days -3 to 180 and taper and mycophenolate mofetil PO three times daily on days 0-28 and then twice daily until day 180 and taper.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Drug: tacrolimus; Drug: mycophenolate mofetil; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation
- Arm II (nontransplant) (Active Comparator): Patients receive mycophenolate mofetil PO twice daily for 16 months, rituximab IV on days 1 and 15 and then repeated at 6 months, and cyclophosphamide IV at 28-32 day intervals or orally once daily for 16 months.
  Interventions: Drug: mycophenolate mofetil; Biological: rituximab; Drug: cyclophosphamide

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
  Arms: Arm I (transplant)
Radiation: total-body irradiation — Undergo total-body irradiation
  Other Names: TBI
  Arms: Arm I (transplant)
Drug: tacrolimus — Given orally
  Other Names: FK 506; Prograf
  Arms: Arm I (transplant)
Drug: mycophenolate mofetil — Given orally
  Other Names: Cellcept; MMF
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
  Arms: Arm II (nontransplant)
Drug: cyclophosphamide — Given orally
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm II (nontransplant)
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo transplantation
  Arms: Arm I (transplant)
Procedure: peripheral blood stem cell transplantation — Undergo transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
  Arms: Arm I (transplant)

SUMMARY:
The purpose of the study is to see how well reduced intensity conditioning followed by a stem cell transplant from a donor (allogeneic) works in treating patients with severe systemic sclerosis. In an allogeneic stem cell transplant procedure, stem cells are taken from a healthy donor and transplanted into the patient. Stem cells can be donated by a family member or an unrelated donor who is a complete tissue type match.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall effects of allogeneic hematopoietic cell transplantation (HCT) in systemic sclerosis (SSc).

II. To assess the potential efficacy, in terms of event-free survival (EFS) at 2 (part 1) and 5 (part 2) years, of allogeneic HCT as treatment for patients with severe SSc.

SECONDARY OBJECTIVES:

I. To evaluate the rate of complications of allogeneic HCT after nonmyeloablative conditioning including the incidence of graft rejection, regimen-related toxicities, severe acute and chronic graft-vs-host disease (GVHD), infectious complications, treatment-related mortality (TRM), and overall survival.

II. To evaluate treatment effects on disease activation/progression, as indicated by measures of cardiac, pulmonary, gastrointestinal and renal function, as well as skin thickness, overall functional assessment (SHAQ), use of concomitant disease-modifying antirheumatic drugs (DMARDs), and occurrence of myositis.

III. To evaluate disease responses after nonmyeloablative conditioning and allogeneic HCT or immunomodulatory therapy, assessing skin disease by modified Rodnan Skin Score (mRSS), pulmonary function as measured by diffusing capacity of the lung for carbon monoxide (DLCO) and forced vital capacity (FVC), Modified Scleroderma Health Assessment Questionnaire (SHAQ), and Quality of Life using Short Form 36 (SF36).

IV. To evaluate, by mechanistic studies, of the effect of allogeneic HCT on dermal fibrosis and vasculopathy.

V. To evaluate the late complications of allogeneic HCT after nonmyeloablative conditioning including the incidence and prevalence of chronic GVHD and time to discontinue immunosuppression, infectious complications, TRM and overall survival.

VI. To evaluate the treatment effects on disease activation/ progression, as indicated by measures of cardiac, pulmonary, gastrointestinal and renal function, as well as skin thickness, overall functional assessment (SHAQ), use of concomitant DMARDs, and occurrence of myositis.

VII. To evaluate disease responses after nonmyeloablative conditioning and allogeneic HCT or immunomodulatory therapy, assessing skin disease by modified Rodnan Skin Score (mRSS), pulmonary function as measured by DLCO and FVC, Modified Scleroderma Health Assessment Questionnaire (SHAQ), and Quality of Life using Short Form 36 (SF36).

OUTLINE: Patients are assigned to 1 of 2 treatment arms and receive nonmyeloablative conditioning followed by an allogeneic peripheral blood stem cell transplantation. Treatment in both arms continues in the absence of disease progression of unacceptable toxicity.

ARM I (transplant): Patients receive fludarabine intravenously (IV) on days -4 to -2. Patients undergo total-body irradiation on day 0. Patients then undergo peripheral blood stem cell transplantation on day 0. Patients receive GVHD prophylaxis comprising tacrolimus orally (PO) twice daily on days -3 to 180 and taper and mycophenolate mofetil PO three times daily on days 0-28 and then twice daily until day 180 and taper.

ARM II (nontransplant): Patients will receive immunosuppressive therapy based on their history. The 3 options that they may receive include 1.)mycophenolate mofetil PO twice daily for 16 months, 2.) Rituximab IV on days 1 and 15 and then repeated at 6 months, and 3.) Cyclophosphamide IV at 28-32 day intervals or orally once daily for 16 months.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe SSc as defined by the American College of Rheumatology and at high-risk for a fatal outcome based on the following prognostic factors from groups 1-5:

   * Group 1: Patients with 1) both a. and b. below; and 2) at least one of c., d. or e:

     * a. Diffuse cutaneous scleroderma with skin score of >= 16 (modified Rodnan skin scale)
     * b. Duration of systemic sclerosis =< 5 years from the onset of first non-Raynaud's symptom
     * c. Presence of interstitial lung disease with FVC or DLCOcorr =< 70% of predicted and evidence of alveolitis (abnormal bronchoalveolar lavage [BAL] or high resolution chest computed tomography [CT] scan)
     * d. Left heart failure with left ventricular ejection Fraction (LVEF) < 50% or pericardial effusion (mild-moderate) or 2nd or 3rd Atrial-Ventricular (AV) block; Myocardial disease not secondary to SSc must be excluded by a cardiologist
     * e. History of SSc-related renal disease that is not active at the time of screening; History of scleroderma hypertensive renal crisis is included in this criterion
   * Group 2: Patients will have progressive pulmonary disease as the primary indication for transplant as defined by a decrease in the FVC or DLCO by 15 percent or greater in the previous 12-month period. In addition, patients may have either less skin involvement than group 1 (mRSS < 16) if they have a history of diffuse cutaneous disease and the FVC or DLCOcorr is < 70% or both FVC and DLCOcorr >= 70% if they have diffuse cutaneous disease (mRSS > 16) at screening for the study; Patients must also have evidence of alveolitis as defined by abnormal chest CT or BAL
   * Group 3: Have progressive active SSc after prior autologous HCT based on the presence of progressive pulmonary disease; This will be defined by a decrease in the FVC since prior autologous transplant by 10 percent or greater, or DLCO since prior autologous transplant by 15 percent or greater in addition to evidence of alveolitis as defined by chest CT changes or BAL; If patients had prior autologous HCT on the SCOT clinical trial, they must have failed based on the defined study endpoints and be approved by the protocol principal investigator (PI)
   * Group 4: Patients who meet group 1 inclusion criteria but have FVC or DLCO < 70% plus have had an adverse event to cyclophosphamide preventing its further use (i.e., hemorrhagic cystitis, leucopenia with WBC, 2000 or ANC < 1000 or platelet count < 100,000 and other adverse events)
   * Group 5: Diffuse scleroderma with disease duration =< 2 years since development of first sign of skin thickening plus modified Rodnan skin score >= 25 plus ESR > 25 mm/1st hour and/or Hb < 11 g/dL not explained by causes other than active scleroderma.
2. Unless patients have a DLCOcorr less than 45%, patients must have failed either oral or intravenous cyclophosphamide regimen defined as:

   * IV cyclophosphamide administration for > 6 months or a total cumulative IV dose of 6 g/m^2, or
   * oral cyclophosphamide administration for > 6 months regardless of dose, or
   * combination of oral and IV cyclophosphamide for > 6 months independent of dose
3. Patient must have a sibling who is a) HLA-identical and b) could serve as a donor of a peripheral blood stem cell graft to be placed on the transplant arm or an unrelated donor matched at HLA-A, B, C, DRB1 and DQB1. Patients without an HLA-identical sibling or an HLA-matched unrelated donor that meet the above criteria will be placed on the non-transplant arm

DONOR:

* The donor must be an HLA-identical sibling of the patient or an HLA-matched unrelated donor.
* If the donor has reached the age of assent, then they must have completed the local institutional review board (IRB) assent process.
* Donor must consent to G-CSF administration and to leukapheresis for HSC collection.
* Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian).
* Age 12-75 years; Pediatric donors must be > 50 kg body weight.

Exclusion Criteria:

* Eligible for the NIH-sponsored randomized clinical trial (SCOT)
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months or until immunosuppression is discontinued following transplantation
* Evidence of ongoing active infection
* Pregnancy
* Subjects with pulmonary, cardiac, hepatic, or renal impairment that would limit their ability to receive therapy and compromise their survival. This includes but is not restricted to, subjects with any of the following:

  * Severe pulmonary dysfunction defined as:

    1. A hemoglobin corrected DLCOcorr < 30% or FVC < 40% of predicted; or
    2. O2 saturation < 92% at rest without supplemental oxygen; or
    3. PO2 < 70 mmHg or pCO2 > 50 mmHg without supplemental oxygen
  * Significant uncontrolled pulmonary hypertension defined as:

    1. Pulmonary artery peak systolic pressure > 45 mmHg by echocardiogram and mean pulmonary artery pressure by right heart catheterization exceeding 32 mmHg at rest or 42 mm Hg during exercise; or
    2. New York Heart Association (NYHA)/World Health Organization (WHO) classification for pulmonary hypertension, Class III or IV
  * Cardiac: Uncontrolled clinically significant arrhythmias; clinical evidence of significant cardiac disease (NYHA Class III or IV); LVEF < 40% by echocardiogram
  * Significant renal pathology, defined as:

    1. Estimated CrCl < 60 mL/min (using Cockcroft-Gault formula based on actual body weight) or serum creatinine > 2.0 mg/dL OR
    2. Active, untreated SSc renal crisis at the time of enrollment
  * Active hepatitis or liver biopsy evidence of cirrhosis or periportal fibrosis. Total bilirubin > 2.5 x the upper limit of normal (and not related to Gilbert's syndrome) and/or Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 4 x the upper limit of normal
  * Patients with poorly controlled hypertension
  * Patients whose life expectancy is severely limited by illness other than autoimmune disease
* DONOR:

  * Identical twin of patient
  * Female donors who are pregnant (positive B-HCG) or breastfeeding
  * Infection with human immunodeficiency virus (HIV) or active viral hepatitis (B or C)
  * Known allergy to G-CSF
  * Current serious systemic illness
  * Uncontrolled bacterial, viral or fungal infection (currently taking medication and progression of clinical symptoms)
  * Donors receiving experimental therapy or investigational agents
  * Donors with cancer other than treated basal cell or carcinoma in situ of cervix; Cancer treated with curative intent > 2 years previous will be reviewed on a case-by-case basis by a Protocol Chair or Medical Monitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | 2 years

SECONDARY OUTCOMES:
Event-free survival | 5 years
Overall survival | 2 years
Overall survival | 5 years
Time to progression | 2 years
Time to progression | 5 years
Incidence of initiation of any SSC disease-modifying therapy other than that specified in the protocol treatment arms | Up to 5 years
Incidence of definite and probable viral, fungal, and bacterial infections | Up to 5 years
Median time to engraftment as defined as having greater than or equal to 5% donor T cells in the peripheral blood (donor T cell chimerism) | From date of transplant to time of engraftment
Rate of primary graft failure | Day 56
Rate of secondary graft failure | 1 year
Probability of acute and chronic GVHD | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: George Georges, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States